CLINICAL TRIAL: NCT02157623
Title: Pilot Trial Comparing Two Different Wavelengths of Light (Blue Versus Red) During Levulan™-Based Photodynamic Therapy of Basal Cell Carcinoma in Patients With Basal Cell Nevus Syndrome
Brief Title: Blue vs Red Light During Levulan Based Photodynamic Therapy in Patients With Basal Cell Nevus Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edward Maytin, MD, PhD (Other)
Collaborators: DUSA Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Edward Maytin, MD, PhD, Staff, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE 2614; NCT02258243 (obsolete NCT alias)
Record Dates: First submitted 2014-06-02; First posted 2014-06-06 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Basal Cell Nevus Syndrome
Keywords: Basal Cell Nevus Syndrome; Gorlin's Syndrome
MeSH Terms: conditions — Basal Cell Nevus Syndrome | interventions — Aminolevulinic Acid; Solutions; Photochemotherapy; Red Light; 1-phenyl-3,3-dimethyltriazene; Blue Light

STUDY DESIGN:
Intervention Model Description: All patients received a different treatment to each half of their body. First Levulan with red light PDT (to tumors on one side of the body), and then Levulan with blue light PDT (to tumors on the other side of the body), at six treatment visits.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Red Light PDT and Blue Light PDT (Experimental): The tumor clearance with one side treated with Levulan and Red light PDT, and the contralateral side treated with Blue light PDT.
  Interventions: Drug: Levulan; Other: Red Light PDT; Other: Blue Light PDT

INTERVENTIONS:
Drug: Levulan — Levulan application followed by Red or Blue light PDT
  Other Names: Levulan™; Levulan® Kerastick® for Topical Solution; 5-aminolevulinic acid; aminolevulinic acid HCL; ALA
Other: Red Light PDT — Aktilite™ (red lamp) after Levulan application on lesions
  Other Names: Aktilite™; Red Lamp; Red Light; PDT
Other: Blue Light PDT — Blu-U® (blue lamp) after Levulan application on lesions
  Other Names: Blu-U; Blue Lamp; Blue Light; PDT

SUMMARY:
The investigators will be testing whether aminolevulinate-based (Levulan™) Photodynamic Therapy (PDT) shows effectiveness in the treatment and prevention of cutaneous basal cell carcinoma (BCC) in Basal Cell Nevus Syndrome (BCNS) patients. Levulan™ PDT is an FDA-approved method widely used currently for squamous precancers of the skin. The investigators hypothesize that PDT will provide exceptional benefit in the BCNS population because PDT is nonmutagenic, nonscarring, and can be safely repeated many times. Additionally, the study will investigate whether there are any differences in tumor clearance between the Blu-U® (blue lamp) and Aktilite™(red lamp) therapies.

DETAILED DESCRIPTION:
This is a pilot intra-patient comparative study to evaluate the ability of cyclic Photodynamic Therapy (PDT) using Red (635 nm) or Blue (400 nm) light with 5-Aminolevulinic acid, to eliminate BCC skin cancers that occur in patients with Basal Cell Nevus Syndrome (Gorlin-Goltz Syndrome).

Patients will receive 3 cycles of Red light and Blue light PDT treatments, for a total of 6 treatments, over a 4 month period. Cycles will be spaced 2 months apart. Each cycle consists of a double course of PDT treatment with treatments spaced one week apart. Every subject will be treated with two light sources, blue and red, according to randomized assignments made to left side or right side of the body. There will be a final assessment visit at month 6.

ELIGIBILITY:
Inclusion Criteria:

* Men, women, and children of any age or ethnic group who meet eligibility
* Patients under 18 years of age must be accompanied and co-consented, by a parent or legal guardian.
* Patients must have a diagnosis of Basal Cell Nevus Syndrome (BCNS)
* For diagnosis of BCNS, the patient must have either 2 major criteria, one major and two minor criteria, or one major criterion plus molecular confirmation of a PTCH1 gene mutation
* Major criteria are:

  * (1) BCC prior to age 20 years, or excessive number of BCCs out of proportion to prior sun exposure and skin type
  * (2) keratocyst of the jaw prior to age 20
  * (3) palmar or plantar pitting
  * (4) lamellar calcification of the falx cerebri
  * (5) medulloblastoma
  * (6) first degree relative with BCNS
* Minor criteria are:

  * (1) rib anomalies, or other specific skeletal malformations including kyphoscoliosis and short 4th metacarpals
  * (2) macrocephaly
  * (3) cleft/lip or palate;
  * (4) fibroma of the heart or ovary
  * (5) ocular abnormalities
  * (6) other rare abnormalities
* At least two BCC tumors, preferably more, located in different body regions or located greater than 10 cm apart in locations that can be reproducibly separated into red and blue illumination fields
* Female subjects are not pregnant or nursing or planning to become pregnant during the study
* Subjects must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Pregnant, planning on getting pregnant or nursing
* Currently participating in another clinical trial
* Using any topical treatment for their BCC tumors, unless discontinued at least 1 month prior
* Currently being treated for other cancers with medical or radiation therapy
* Patients with a known hypersensitivity to 5-aminolevulinic acid or any component of the study material
* Patients with a history of a photosensitivity disease, including porphyria cutanea tarda

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward V. Maytin, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Red Light/Blue Light Participants: Subjects will receive Red Light PDT on one side of the body, and Blue Light PDT to the contralateral side.
Period: Overall Study
Arm/Group | Red Light/Blue Light Participants
Started | 3 (3 patients, each received red light on half of body and blue light on the contralateral side.)
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Red Light / Blue Light Participants: Subject will be receive red light PDT on one side of the body, and blue light PDT to the contralateral side after Levulan application
Arm/Group | Red Light / Blue Light Participants
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 42 [33 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Tumor Clearance Rate Following Red or Blue Light PDT
Description: The rate of clearance of existing BCC tumors will be assessed in patients with BCNS, using clinical and photographic measurements. The endpoint will be assessed for tumors in a Red light treatment field and a Blue light treatment field in each patient, and compared (bilateral intrapatient comparison).
Time Frame: 6 months
Population: Three (3) patients with BCNS were enrolled.
Measure: Mean (Full Range); unit: Percentage of tumors cleared
Units Other Than Participants: Tumors
Groups:
- Red Light Photodynamic Therapy: One side of patient received red light PDT
- Blue Light Photodynamic Therapy: The other side of the patient received blue light PDT
Arm/Group | Red Light Photodynamic Therapy | Blue Light Photodynamic Therapy
Number analyzed (Participants) | 3 | 3
Number analyzed (Tumors) | 76 | 65
Percentage of tumors cleared | 87.3 [75 to 96] | 99 [97 to 100]

2. Secondary Outcome: Pain During Illumination
Description: Pain reported by the patient, using a 0-10 Visual Analog Scale (VAS), where 0 is no pain and 10 is maximum pain possible.
Time Frame: Maximum value reported during the illumination period
Measure: Mean (Standard Error); unit: VAS score value
Groups:
- Pain During Red Light: Pain during red light illumination (on a 0-10 visual analog scale)
- Pain During Blue Light: Pain during blue light illumination (on a 0-10 visual analog scale)
Arm/Group | Pain During Red Light | Pain During Blue Light
Number analyzed (Participants) | 3 | 3
VAS score value | 5.6 (2.0) | 3.7 (1.7)

3. Secondary Outcome: Patient Satisfaction Survey
Description: Overall patient satisfaction with the technique will be assessed using a simple survey:
  6 = extremely satisfied; 5 = very satisfied; 4 = somewhat satisfied; 3 = somewhat dissatisfied; 2 = very dissatisfied; 1 = extremely dissatisfied.
Time Frame: 6 months
Measure: Mean (Full Range); unit: Scores on the rating scale
Groups:
- Red Light Treatment: RATING SCALE: 6 = extremely satisfied; 5 = very satisfied; 4 = somewhat satisfied; 3 = somewhat dissatisfied; 2 = very dissatisfied; 1 = extremely dissatisfied.
- Blue Light Treatment: 1 to 6 satisfaction scale
Arm/Group | Red Light Treatment | Blue Light Treatment
Number analyzed (Participants) | 3 | 3
Scores on the rating scale | 5.3 [5 to 6] | 5.6 [5 to 6]

ADVERSE EVENTS:
Groups:
- Red Light Photodynamic Therapy: Subject will be randomized to right or left side and assigned side will be treated with red light PDT after Levulan application
  Levulan: Levulan application followed by Red or Blue light PDT on randomized treatment fields
  Red Light Photodynamic Therapy: Aktilite™ (red lamp) after Levulan application on randomized treatment field
- Blue Light Photodynamic Therapy: Subject will be randomized to right or left side and assigned side will be treated with blue light PDT after Levulan application
  Levulan: Levulan application followed by Red or Blue light PDT on randomized treatment fields
  Blue Light Photodynamic Therapy: Blu-U® (blue lamp) after Levulan application on randomized treatment field
Arm/Group | Red Light Photodynamic Therapy | Blue Light Photodynamic Therapy
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes